CLINICAL TRIAL: NCT00767481
Title: 1 Year Study Trav/Brinz QD Fixed Combination Versus COSOPT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Project Cancelled
Sponsor: Alcon Research (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-08-16; 2008-002781-66
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2011-11

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: glaucoma; Patients with open-angle glaucoma or ocular hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Travoprost; brinzolamide; dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Travoprost/Brinzolamide PM, Vehicle AM (Experimental): Travoprost/Brinzolamide PM, Vehicle AM
  Interventions: Drug: Travoprost/Brinzolamide
- Travoprost/Brinzolamide AM, Vehicle PM (Experimental): Travoprost/Brinzolamide AM, Vehicle PM
  Interventions: Drug: Travoprost/Brinzolamide
- Cosopt (Active Comparator): Cosopt BID
  Interventions: Drug: Cosopt

INTERVENTIONS:
Drug: Travoprost/Brinzolamide — Eye drop suspension, once daily
  Arms: Travoprost/Brinzolamide AM, Vehicle PM; Travoprost/Brinzolamide PM, Vehicle AM
Drug: Cosopt — Eye drop solution, one drop BID
  Arms: Cosopt

SUMMARY:
Parallel, Multi-Center, Double-masked, Active controlled, three arm study comparing the IOP lowering efficacy and safety over 12 months of morning or evening instillations of Travoprost/Brinzolamide vs. Cosopt dosed in the morning and evening in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* IOP at screening visit <18mmHg in at least one eye Mean IOP in same eye (at both eligibility 1 &2 visits)

  * 24 and ≤ 36 mmHg at 9:00
  * 21 and ≤ 36 mmHg at 11:00 and 16:00

Exclusion Criteria:

* Severe central visual field loss Angle Shaffer grade < 2 C/D ratio > 0.8 (horizontal or vertical measurement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Mean IOP | 9:00,11:00, and 1600 time points at month 12

SECONDARY OUTCOMES:
Percent change in IOP, IOP change from baseline, patients with IOP <18mmHg. BSCVA, Ocular signs, Dilated fundus, perimetry, pachymetry, cardiovascular parameters(pulse, BP and AEs at W2, W3, M6, M9 and M12. | All on therapy time points not included in primary efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Mexico City, Mexico